CLINICAL TRIAL: NCT00000772
Title: A Phase I Open-Label Study of the Safety, Tolerance, and Pharmacokinetic Interactions of Combination Didanosine and Ribavirin in HIV-Positive Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); ICN Pharmaceuticals (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 231; 11208 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Ribavirin; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ribavirin; Didanosine

INTERVENTIONS:
Drug: Ribavirin
Drug: Didanosine

SUMMARY:
To evaluate the safety and tolerance of concurrent administration of standard-dose didanosine (ddI) with low-dose ribavirin in HIV-positive patients. To determine the pharmacokinetic interactions of concurrent administration of ddI and ribavirin and correlate pharmacokinetic parameters with toxicity. To investigate antiviral activity of the combined regimen.

Combination ddI/ribavirin therapy, if safe and effective, offers an alternative combination antiretroviral regimen for patients unable to tolerate regimens containing zidovudine (AZT).

DETAILED DESCRIPTION:
Combination ddI/ribavirin therapy, if safe and effective, offers an alternative combination antiretroviral regimen for patients unable to tolerate regimens containing zidovudine (AZT).

Patients receive ddI alone for 4 weeks, followed by 8 weeks of combination ddI/ribavirin. Patients who complete the first 12 weeks without major toxicity may receive an additional 12 weeks of combination therapy on an optional basis. Patients are followed for 60 days after the last treatment visit.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Stable maintenance or prophylaxis therapy for opportunistic infection, if such therapy was administered for at least 30 days prior to study entry.
* Isoniazid for chemoprophylaxis against Mycobacterium tuberculosis.
* Fluconazole for mucosal candidiasis or cryptococcosis.
* Acyclovir (up to 1.0 g/day).
* Dapsone.
* Ketoconazole.
* Quinolones.
* Tetracycline.
* Vitamins and herbal therapies.
* Antibiotics as clinically indicated.
* Systemic corticosteroids for < 21 days for acute problems.
* Regularly prescribed medications.

Patients must have:

* HIV positivity by ELISA confirmed by Western blot.
* CD4 count < 500 cells/mm3 within 30 days prior to study entry.
* No active opportunistic infections requiring treatment (patients on stable maintenance and prophylaxis therapy for opportunistic infections for at least 30 days are permitted).

NOTE:

* Enrollment of women is encouraged.

Prior Medication:

Allowed:

* Prior stable maintenance or prophylaxis therapy for opportunistic infection, if administered for at least 30 days prior to study entry.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Concurrent rifampin or rifabutin.
* Other anti-HIV drugs and investigational agents.
* Biological response modifiers.
* Ganciclovir or foscarnet.
* Systemic cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Concurrent radiation therapy other than limited localized therapy to the skin.

Patients with the following prior conditions are excluded:

* History of peripheral neuropathy.
* History of pancreatitis or active liver disease.

Prior Medication:

Excluded:

* Prior ddI.
* Ribavirin within 60 days prior to study entry.
* AZT or ddC within 2 weeks prior to study entry.

Prior Treatment:

Excluded:

* Transfusion within 2 weeks prior to study entry.

Active alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Japour AJ, Study Chair; Lertora JJ, Study Chair; Crumpacker C, Study Chair
Locations (2):
- United States (2):
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota

REFERENCES:
- [Background] Japour AJ, et al. A Phase I study of the safety, tolerance, & pharmacokinetics of combination didanosine/ribavirin for HIV disease (ACTG 231). Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:103